CLINICAL TRIAL: NCT04364399
Title: Randomized, Double-blind, Controlled Phase Ⅳ Clinical Trial to Evaluate the Safety and Immunogenicity of Mumps Vaccine in Healthy Infants Aged 8 ~12 Months.
Brief Title: Clinical Trial to Evaluate the Safety and Immunogenicity of Mumps Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-MUMPS-4006
Record Dates: First submitted 2020-04-07; First posted 2020-04-28 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Mumps
Keywords: Mumps; Mumps vaccine; measles, mumps and rubella combined vaccine, live; infants
MeSH Terms: conditions — Mumps; Measles | interventions — Mumps Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Mumps vaccine, one dose
  Interventions: Biological: Mumps vaccine
- Control group (Active Comparator): measles, mumps and rubella combined vaccine, live, one dose
  Interventions: Biological: measles, mumps and rubella combined vaccine, live

INTERVENTIONS:
Biological: Mumps vaccine — One dose of mumps vaccine: 0.5 ml per dose, mumps live virus not less than 3.7 lg CCID50
  Arms: Experimental group
Biological: measles, mumps and rubella combined vaccine, live — One dose of measles, mumps and rubella combined vaccine, live: 0.5 ml per dose, mumps live virus not less than 4.3 lg CCID50
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of mumps vaccine in healthy infants aged 8-12months, compared with measles, mumps and rubella combined vaccine, live (MMRV).

DETAILED DESCRIPTION:
The study is a randomized, double-blind, controlled phase Ⅳ clinical trial. And 920 infants will be assigned to investigational group and controlled group in a 1:1 ratio. The investigational vaccine is manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd. The controlled vaccine is manufactured by Shanghai institute of biological products Co., Ltd.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 8 - 12 months old;
* Proven legal identity;
* Written consent of the guardian(s) of the volunteer

Exclusion Criteria:

* Received mumps vaccine or vaccine containing mumps virus;
* History of mumps;
* Axillary temperature > 37.4 °C;
* History of allergy to any vaccine or vaccine ingredient;
* History of serious adverse reaction(s) to vaccination, such as urticaria, difficulty in breathing, angioneurotic edema, abdominal pain, etc;
* Autoimmune disease or immunodeficiency or immunosuppression;
* Congenital malformation, genetic defects, severe malnutrition;
* Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities) , or obvious bruising or coagulation disorders;
* Severe chronic diseases (e.g., severe cardiovascular disease, liver and kidney disease beyond the control of drugs, or cancer)
* Severe neurological disorders (epilepsy, seizures or convulsions) or psychosis;
* History of thyroidectomy, absence of spleen, functional absence of spleen, and any condition resulting from absence of spleen or splenectomy;
* Receipt of any of the following products:

  1. Any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
  2. Any live attenuated vaccine within 28 days prior to study entry;
  3. Any other investigational medicine(s) or vaccine within 30 days prior to study entry;
  4. Blood product within 3 months prior to study entry;
  5. Any immunosuppressant, cytotoxic medicine, or oral corticosteroids;
  6. Any of the acute disease or attack of the chronic disease within 7 days;
  7. Pregnant in cohabitants or congenital immune diseases;
  8. Based on the judgment of investigator(s), there was any condition indicating that the subject should be excluded

Ages: 8 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 920 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
The seroconversion rate of hemagglutination inhibition (HI) antibody | the 30th day after vaccination
  Immunogenicity index, One of the standard to evaluate the immunogenicity of experimental vaccine

SECONDARY OUTCOMES:
The GMT of HI antibody | the 30th day after vaccination
  Immunogenicity index, Another standard to evaluate the immunogenicity of experimental vaccine
The incidence of the solicited local and systemic adverse reactions | from day 0 to day 14 after vaccination
  Safety index, The adverse reactions refers to the adverse events which were considered related to the vaccination
The incidence of the unsolicited adverse events | from day 0 to day 30 after immunization
  Safety Index
The incidence of the serious adverse events | from day 0 to day 30 after immunization
  Safety Index

CONTACTS AND LOCATIONS:
Overall Officials: Lirong Huang, Bachelor, Principal Investigator — Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control
Locations (1):
- Hezhou Center for Disease Prevention and Control, Hezhou, Guangxi, China

IPD SHARING:
Plan to Share IPD: No